CLINICAL TRIAL: NCT06179225
Title: Reducing Loneliness of Older Adults in Long Term Care Facilities Through Collaborative Augmented Realities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Nilanjan Sarkar, Professor, Mechanical Engineering, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 078480; R21AG078480 (NIH)
Record Dates: First submitted 2023-12-02; First posted 2023-12-21 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Loneliness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HMD AR (Experimental): Pairs of older adults with their designated family members who geographically apart will perform collaborative activities using HMD AR in 8 sessions over 4 weeks.
  Interventions: Behavioral: HMD AR
- 2-D Audio-Visual (Active Comparator): Pairs of older adults with their designated family members who geographically apart will perform collaborative activities using 2-D Audio-Visual in 8 sessions over 4 weeks.
  Interventions: Behavioral: 2-D AV

INTERVENTIONS:
Behavioral: HMD AR — Older adults will wear head mounted display to engage in collaborative augmented reality activities: sharing a meal, playing board games, and decorating home.
  Arms: HMD AR
Behavioral: 2-D AV — Older adults will use 2-D AV to engage with family members at a distance.
  Arms: 2-D Audio-Visual

SUMMARY:
The goal of this clinical trial is to test the use of head-mounted display (HMD) augmented reality (AR) in older adults residing in long term care communities. The main questions it aims to answer are: what is the feasibility, acceptability, and satisfaction of HMD AR vs two-dimensional audio-video communication? Older adults and their designated family member will complete HMD AR activities in 8 session visits over 4 weeks. Researchers will compare HMD AR to 2-D audio-visual (AV) comparison group on feasibility, acceptability, and satisfaction with the interactive communication technology.

DETAILED DESCRIPTION:
For both interventions, the bandwidth within the family members' homes will be measured and a hotspot created if necessary to facilitate data streaming. For each session, a trained research assistant (RA) will be physically present at the Long-term Care (LTC) to troubleshoot for technological issues. The RA will observe the staff member establish the Interactive Communication technology (ICT) connection between the older adult and family member, assisting as needed. The RA and staff member will remain within the room; the RA will monitor for technological issues. The staff member will monitor the older adults' reactions.

HMD-AR Intervention Experimental Setup. For the older adults, equipment set-up will be in a dedicated room at the LTC that allows for environmental overlays. Equipment includes two Kinect cameras, one HMD and one E4 wrist sensor that the older adult will wear to measure stress through physiological sensing. The family member will be consulted for placement of the 2 Kinect cameras in their home.

AR Activities. At least one meal session and one activity session will be conducted. The remaining sessions will consist of activities based on the preference of the older adult-family member. Staff will be trained to turn on the headset, computers, and ensure communication connection between the older adult and family member.

2D Audio-visual Intervention The 2D audio-visual sessions will take place in a dedicated room at the LTC. Staff will initiate the connection between the older adult and family member. In the unlikely event a family member does not have a device for the 2D audio-visual visits, a computer tablet will be supplied for use during the study.

ELIGIBILITY:
Inclusion Criteria:

* age 60 and older
* residing at LTC greater than 3 months

Exclusion Criteria:

* unable to provide assent or consent
* unable to understand or speak English
* physical impairment that impedes participation
* terminally ill

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure (FIM) questionnaire | Week 4
  questionnaire
Acceptability of Intervention Measure (AIM) | Week 4
  The degree to which the technology is acceptable to older adults and their family members.
UCLA Loneliness Scale | Baseline and week 4
  Measure of loneliness of older adults
Networked Minds Measure (NMM) of Social Presence | Week 4
  Measure of Social Presence, which is the psychological phenomenon in which others are perceived as physical 'real' persons in ICT

CONTACTS AND LOCATIONS:
Overall Officials: Nilanjan Sarkar, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified data will be provided upon request.

DOCUMENTS (1):
  • Informed Consent Form (2024-11-11): https://cdn.clinicaltrials.gov/large-docs/25/NCT06179225/ICF_000.pdf